CLINICAL TRIAL: NCT07400185
Title: Evaluation Of The Effects Of Changes In Operating Table Position On Perfusion Index And Spinal Anesthesia: An Observational Study
Brief Title: Evaluation Of The Effects Of Changes In Operating Table Position On Perfusion Index And Spinal Anesthesia
Acronym: Perfusion
Status: Not yet recruiting | Type: Observational
Sponsor: Enes Celik (Other)
Responsible Party: Sponsor-Investigator, Enes Celik, ANESTHESIOLOGIST, Mardin Artuklu University
Organization: Mardin Artuklu University (Other)
Other Study IDs: 26.12.2025-2-01
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Perfusion Index; Position Differences
Keywords: The Effects of Changes in Operating Table Position on Perfusion Index and Spinal Anesthesia; operating table position

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neutral group: Patients will be included who are positioned so that the operating table is neutral.
- tilt group: Patients will be positioned on the operating table with an incline towards the side they will be operated on.

SUMMARY:
The aim of this observational study is to investigate how table position affects the development of block in patients undergoing spinal anesthesia. Perfusion index measurements will be used to answer this question. Patients who will undergo perfusion index measurement during surgery will be included in the study. These patients will be compared with patients whose anesthesiologists chose not to position them on the operating table. The study is planned to continue for approximately 40 days, and the data collected during this period will be used for evaluation.

DETAILED DESCRIPTION:
Patients aged 18-65 years in ASA1-3 risk group who will undergo lower extremity surgery with spinal anesthesia are planned to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo lower extremity surgery within the specified time frame, are in ASA 1-3 risk group, have no additional medical conditions, and will receive spinal anesthesia.

Exclusion Criteria:

* Patients under 18 and over 65 years of age Patients who have received anesthesia other than spinal anesthesia Patients with peripheral artery disease Patients with nail polish, etc. on their nails

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo lower extremity surgery within the specified time frame, are in ASA 1-3 risk group, have no additional medical conditions, and will receive spinal anesthesia.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
perfusion index | 5 min
  The amount of increase over time will be recorded according to the basal perfusion index value.

CONTACTS AND LOCATIONS:
Locations (1):
- Mardin Artuklu University Training and Research Hospital, Mardin, Artuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
In accordance with the personal data protection law, personal data may be shared for scientific purposes after being anonymized.

REFERENCES:
- [Background] Tapar H, Karaman S, Dogru S, Karaman T, Sahin A, Tapar GG, Altiparmak F, Suren M. The effect of patient positions on perfusion index. BMC Anesthesiol. 2018 Aug 17;18(1):111. doi: 10.1186/s12871-018-0571-z. PMID 30115011